CLINICAL TRIAL: NCT02132832
Title: Buspirone, Stress, and Attentional Bias to Marijuana Cues
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Scott Lane, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: buspirone, stress, marijuana; R21DA034825 (NIH)
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Cannabis Use Disorder
Keywords: marijuana; attentional bias; stress; buspirone
MeSH Terms: conditions — Marijuana Abuse | interventions — Buspirone; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buspirone (Experimental): Buspirone is administered orally twice per day (9:00 AM and 6:00 PM) for 3 weeks. 10 mg buspirone is administered on days 1-4, then the dose is increased by 10 mg every 3 days to a maximum of 40 mg buspirone on days 10-19.
  Interventions: Drug: Buspirone
- Placebo (Placebo Comparator): Placebo is administered orally twice per day (9:00 AM and 6:00 PM) for 3 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone — Buspirone is an anxiolytic compound marked by modulation of both 5-HT1A and D3 receptors. Buspirone is administered orally twice per day (9:00 AM and 6:00 PM) for 3 weeks. 10 mg buspirone is administered on days 1-4, then the dose is increased by 10 mg every 3 days to a maximum of 40 mg buspirone on days 10-19.
  Arms: Buspirone
Drug: Placebo — Placebo is administered orally twice per day (9:00 AM and 6:00 PM) for 3 weeks.
  Other Names: corn starch
  Arms: Placebo

SUMMARY:
This project has two primary goals. The first goal is to further scientific understanding about marijuana abuse by examining two recognized factors in marijuana use and relapse: (1) stress/anxiety and (2) atypical reactivity to marijuana-related stimuli (e.g., attentional bias). The second goal is to attenuate the influence of stress/anxiety and attentional bias to marijuana stimuli via administration of buspirone.

Buspirone is uniquely suited to this project because it has effects on neurotransmitter systems known to modulate both stress/anxiety and attentional bias.

DETAILED DESCRIPTION:
For nearly 40 years marijuana has remained the most widely used illicit drug in the US, with more than 50% of first-time users < age 18. Marijuana accounts for ≈ 60% of illicit substance use disorders (SUD) in the US, bearing by percent the largest US public health burden among illicit substances. Across preclinical, human laboratory, and clinical interview data, there is compelling evidence that the phenomenon of cue reactivity is related to drug seeking and relapse. Attentional bias is a measurable component of cue reactivity, and can be operationally defined as differential attention (e.g., reaction time difference) towards drug-related stimuli vs. neutral stimuli. This phenomenon has been demonstrated in SUD populations across many classes of abused drugs, including alcohol, nicotine, stimulants, opiates, and - importantly - marijuana. Cue reactivity and attentional bias are exacerbated by acute and chronic stress and anxiety. Notably, stress is a well-documented predictor of marijuana abuse and marijuana relapse. Therapeutic interventions that attenuate attentional bias to marijuana cues are a potentially important component in the treatment of marijuana SUD. Due to the well-documented association with stress, an intervention that simultaneously addresses both stress and attentional bias could be uniquely efficacious. Currently, few pharmacotherapies exist for marijuana SUD, and none are presently known to address attentional bias to marijuana cues. This application will explore the potential of the anxiolytic buspirone to modify attentional bias and stress. Buspirone is a unique compound marked by modulation of both serotonin (5-HT1A) and dopamine D3 receptors. Importantly, the 5-HT1A receptor is known to play a key role in stress related anxiety, and preclinical work indicates that D3 antagonists significantly decrease cue reactivity to a number of abused drugs. This combination of effects suggests buspirone may be advantageous in targeting both stress and attentional bias as factors that contribute to problem marijuana use.

Accordingly, this project seeks to examine the effects of chronic buspirone administration on attentional bias and stress/anxiety in marijuana SUD. Using laboratory-based methodologies sensitive to attentional bias towards marijuana cues and well validated measures of stress and anxiety, we will examine if buspirone's unique mechanism of action will (a) produce an attenuation of attentional bias to marijuana cues, and (b) be most pronounced under conditions in which attentional bias is related to high levels of stress and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Marijuana substance use disorder based on a score of ≥ 13 on the Cannabis Use Disorders Identification Test - Revised (CUDIT-R)
* a score of ≥ 4 on the Cannabis Abuse Screening Test (CAST)
* meeting criteria for a marijuana substance use disorder based on the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV)

Exclusion Criteria:

* Current DSM-IV Axis I disorder other than marijuana use disorder
* serious medical illness requiring ongoing medical treatment, which could affect the central nervous system, or any other medical contraindication (e.g., renal, cardiovascular, pulmonary, blood) as determined by medical screening
* a positive pregnancy test or breast feeding (females)
* concomitant use of prescription medications that could affect the central nervous system
* active suicidal ideation or Beck Depression Inventory II score greater than 19
* positive urine drug screen for drugs other than marijuana or positive breath alcohol screen
* Shipley-2 test of cognitive aptitude score outside 2 SD units of the published composite score average
* smoking > 10 nicotine cigarettes per day / Fagerstrom Score > 4
* taking meds known to have significant drug interactions with buspirone.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D. Lane, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center - Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 45 were enrolled (i.e., screened and consented), but 3 participants never returned to begin the study. Thus, only 42 participants began the study.
Period: Overall Study
Arm/Group | Buspirone | Placebo
Started | 19 | 23
Completed | 16 | 16
Not Completed | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buspirone | Placebo | Total
Number analyzed (Participants) | 19 | 23 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.16 (7.15) | 29.52 (6.89) | 29.34 (7.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 11 | 13 | 24
Region of Enrollment [Number; unit: participants]
  United States | 19 | 23 | 42

OUTCOME MEASURES:

1. Primary Outcome: Attentional Bias to Marijuana Specific Stimuli Measured Via Analysis of Eye Movements
Description: Eye movements are analyzed using a MiraMetrix S2 Eyetracker. This outcome measure reports a ratio: [(number of anti-saccade errors with marijuana-related images) divided by (total number of anti-saccade errors with marijuana-related images or neutral images)]. Anti-saccade errors are when the subject fails to inhibit fixation onto the image.
Time Frame: week 1
Measure: Mean (Standard Deviation); unit: ratio of errors (see OM description)
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 16 | 16
ratio of errors (see OM description) | 0.5795019 (0.1609511) | 0.5539831 (0.1442601)

2. Primary Outcome: Attentional Bias to Marijuana Specific Stimuli Measured Via Analysis of Eye Movements
Description: as for outcome 1
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: ratio of errors (see OM description)
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 16 | 16
ratio of errors (see OM description) | 0.5517691 (0.1319968) | 0.4979594 (0.1486691)

3. Primary Outcome: Attentional Bias to Marijuana Specific Stimuli Measured Via Analysis of Eye Movements
Description: as for outcome 1
Time Frame: week 3
Measure: Mean (Standard Deviation); unit: ratio of errors (see OM description)
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 16 | 16
ratio of errors (see OM description) | 0.5503957 (0.1133407) | 0.531073 (0.1991689)

4. Primary Outcome: Stress as Assessed by the Perceived Stress Scale
Description: The Perceived Stress Scale is a 10 item scale that was developed to measure the degree to which individuals appraise their life as stressful and has been widely used in health studies. The scale has a 5-point Likert response format. The total score is calculated by summing responses. The questions are general in nature and relatively content free with regard to specific population groups. The range of scores is 0-40, with 40 indicating the most stress.
Time Frame: week 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 16 | 16
units on a scale | 15.05556 (5.885898) | 18.57895 (6.551639)

5. Primary Outcome: Stress as Assessed by the Perceived Stress Scale
Description: as for outcome 4
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 16 | 16
units on a scale | 13.88889 (6.434182) | 16.42105 (5.708822)

6. Primary Outcome: Stress as Assessed by the Perceived Stress Scale
Description: as for outcome 4
Time Frame: week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 16 | 16
units on a scale | 10.38889 (6.436467) | 14.05263 (7.799385)

7. Primary Outcome: Anxiety as Assessed by the Zung Self-Rated Anxiety Scale
Description: The Zung Self-Rated Anxiety Scale is a widely-used 20 item scale that is scored on a Likert-type scale of 1-4, with 15 questions concerning increasing anxiety levels and five questions concerning decreasing anxiety levels. The scale focuses on the most common general anxiety symptoms and means of coping with stressors that produce anxiety. The range of scores is 20-80:
  * 20-44 Normal Range
  * 45-59 Mild to Moderate Anxiety Levels
  * 60-74 Marked to Severe Anxiety Levels
  * 75-80 Extreme Anxiety Levels
Time Frame: week 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 16 | 16
units on a scale | 32.44444 (2.955) | 32.52632 (4.880442)

8. Primary Outcome: Anxiety as Assessed by the Zung Self-Rated Anxiety Scale
Description: as for outcome 7
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 16 | 16
units on a scale | 31.5 (3.714043) | 31.57895 (3.79057)

9. Primary Outcome: Anxiety as Assessed by the Zung Self-Rated Anxiety Scale
Description: as for outcome 7
Time Frame: week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 16 | 16
units on a scale | 33.27778 (4.884616) | 31.63158 (4.125941)

10. Primary Outcome: Stress as Assessed by the Visual Analogue Stress Scale-Current (VASS-C)
Description: With the Visual Analogue Stress Scale - Current (VASS-C), current stress level is ranked on a 0 - 10 visual analog scale, with 0 as no stress and 10 as extreme stress, cued by the question "Please rate your current stress level."
Time Frame: week 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 16 | 16
units on a scale | 3.888889 (2.373602) | 3.631579 (3.515213)

11. Primary Outcome: Stress as Assessed by the Visual Analogue Stress Scale-Current (VASS-C)
Description: as for outcome 10
Time Frame: week 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 16 | 16
units on a scale | 3 (2.44949) | 2.789474 (2.636895)

12. Primary Outcome: Stress as Assessed by the Visual Analogue Stress Scale-Current (VASS-C)
Description: as for outcome 10
Time Frame: week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buspirone | Placebo
Number analyzed (Participants) | 16 | 16
units on a scale | 1.944444 (1.862074) | 2.526316 (2.50263)

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: National Institute on Drug Abuse (NIDA) Serious Adverse Event Tracking and Reporting System (SAETRS); side effects profile
Arm/Group | Buspirone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/23
Other Adverse Events (participants affected / at risk) | 1/19 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buspirone (N=19) | Placebo (N=23)
light-headed, dizziness (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study intends to evaluate reduction of attentional-bias in non-treatment seekers, and it is not designed or powered to address treatment effects on marijuana use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes